CLINICAL TRIAL: NCT02023658
Title: Systems Analysis and Improvement to Optimize pMTCT: A Cluster Randomized Trial
Brief Title: Systems Analysis and Improvement to Optimize pMTCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Network of AIDS Researchers of Eastern and Southern Africa (Unknown); Centro de Investigacao Operacional da Beira (Unknown); Health Alliance International (Other); Eduardo Mondlane University (Other)
Responsible Party: Principal Investigator, Kenneth Sherr, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 44167-EG; R01HD075057 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-30 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: HIV
Keywords: HIV; pMTCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systems analysis and improvement (Experimental): pMTCT systems analysis and improvement
  Interventions: Other: pMTCT systems analysis and improvement
- Control (No Intervention): No systems analysis and improvement intervention for prevention of mother to child HIV transmission services in place.

INTERVENTIONS:
Other: pMTCT systems analysis and improvement — Five-step systems analysis and iterative improvement cycles carried out over a six-month period in intervention facilities.
  Arms: Systems analysis and improvement

SUMMARY:
Despite significant increases in global health investment and the availability of low-cost, efficacious interventions designed to reduce mother to child HIV transmission in low and middle income countries with high HIV burden, the translation of these scientific advances into effective delivery strategies has been slow, uneven and incomplete. As a result, pediatric HIV infection remains largely uncontrolled. Enhancing the implementation of pMTCT interventions through contextually appropriate systems analysis and improvement approaches can potentially reduce drop-offs along the pMTCT cascade, leading to dramatic improvements in infant and maternal outcomes. The goal of this proposal is to develop a model for systematic assessment and improvement of pMTCT services in sub-Saharan Africa. In specific aim 1, we will identify health system factors and service delivery approaches associated with high and low performing pMTCT services in Côte d'Ivoire, Kenya and Mozambique. In specific aim 2 we will adapt evaluate the feasibility and impact of a systems analysis tool and associated performance enhancement approach for pMTCT services in Côte d'Ivoire, Kenya and Mozambique. This systems analysis tool and associated performance enhancement approach is currently being developed and piloted for pMTCT services in Mozambique. The results of this implementation research are expected to generate knowledge of global health significance, and by disseminating the study results and intervention tools through the broad PEPFAR network, can rapidly impact pMTCT service delivery enhancements across the highest need countries.

ELIGIBILITY:
Inclusion Criteria:

* health facility with pMTCT services in central Mozambique, northern Cote d'Ivoire or western Kenya
* health facility with at least 20 HIV-infected women identified in antenatal care per year

Exclusion Criteria:

* health facility over 20 kilometers from a main transport corridor
* health facility with an ongoing prospective study or systems analysis and improvement approach in place

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Uptake of HIV counseling and testing at first antenatal care visit | Patients will be assessed at first antenatal care visit (average of 25 weeks gestational age)
  # women counseled and tested for HIV in their first ANC visit/# first ANC visits
Uptake of CD4 testing at antenatal care | Patients will be assessed during the antenatal care period (average of 25-40 weeks gestational age)
  # CD4 counts of HIV-infected pregnant women/# HIV-infected women newly identified in ANC
Use of appropriate ARVs in pregnancy for prophylaxis or initiation of ART during pregnancy | Patients will be assessed during the antenatal care period (average of 25-40 weeks gestational age)
  # HIV-infected pregnant women starting AZT prophylaxis or ART /# women testing HIV-positive in ANC 3 months previously
Infant HIV determination | 6 weeks post-partum
  # infants <6 weeks of age receiving a PCR test/# women testing HIV-positive in ANC 5 months previously

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Sherr, PhD, Principal Investigator — University of Washington
Locations (3):
- Ministry of Health, Bouaké, Côte d’Ivoire
- Ministry of Health, Nairobi, Kenya
- Ministry of Health, Beira, Sofala, Mozambique

REFERENCES:
- [Background] Sherr K, Gimbel S, Rustagi A, Nduati R, Cuembelo F, Farquhar C, Wasserheit J, Gloyd S; With input from the SAIA Study Team. Systems analysis and improvement to optimize pMTCT (SAIA): a cluster randomized trial. Implement Sci. 2014 May 8;9:55. doi: 10.1186/1748-5908-9-55. PMID 24885976
- [Result] Gimbel S, Rustagi AS, Robinson J, Kouyate S, Coutinho J, Nduati R, Pfeiffer J, Gloyd S, Sherr K, Granato SA, Kone A, Cruz E, Manuel JL, Zucule J, Napua M, Mbatia G, Wariua G, Maina M; with input from the SAIA study team. Evaluation of a Systems Analysis and Improvement Approach to Optimize Prevention of Mother-To-Child Transmission of HIV Using the Consolidated Framework for Implementation Research. J Acquir Immune Defic Syndr. 2016 Aug 1;72 Suppl 2(Suppl 2):S108-16. doi: 10.1097/QAI.0000000000001055. PMID 27355497
- [Derived] Rustagi AS, Gimbel S, Nduati R, Cuembelo Mde F, Wasserheit JN, Farquhar C, Gloyd S, Sherr K; with input from the SAIA Study Team. Implementation and Operational Research: Impact of a Systems Engineering Intervention on PMTCT Service Delivery in Cote d'Ivoire, Kenya, Mozambique: A Cluster Randomized Trial. J Acquir Immune Defic Syndr. 2016 Jul 1;72(3):e68-76. doi: 10.1097/QAI.0000000000001023. PMID 27082507
- [Derived] Gimbel S, Voss J, Mercer MA, Zierler B, Gloyd S, Coutinho Mde J, Floriano F, Cuembelo Mde F, Einberg J, Sherr K. The prevention of mother-to-child transmission of HIV cascade analysis tool: supporting health managers to improve facility-level service delivery. BMC Res Notes. 2014 Oct 21;7:743. doi: 10.1186/1756-0500-7-743. PMID 25335783